CLINICAL TRIAL: NCT03624972
Title: Enhancing Patient-Provider Communication About Sexual Concerns in Breast Cancer: Patient Intervention Study
Brief Title: Addressing Sexual Concerns in Breast Cancer: Patient Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-833-02
Record Dates: First submitted 2018-07-20; First posted 2018-08-10 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer Female
Keywords: communication; sexual health; menopausal health
MeSH Terms: conditions — Communication | interventions — Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resources Only (Active Comparator): Patients will receive a list of resources on sexual and menopausal health in breast cancer. They will be asked to review the resources before their next clinic visit.
  Interventions: Behavioral: Sexual and Menopausal Health Resources
- Resources + Video (Experimental): Patients will receive a list of web resources on sexual and menopausal health in breast cancer. In addition to the resources, patients will be asked to view an online video called "Starting the Conversation" and to complete an accompanying workbook. Patients in this arm will be asked to review the resource list, watch the Starting the Conversation video, and complete the workbook before their next clinic visit.
  Interventions: Behavioral: Starting the Conversation Video; Behavioral: Sexual and Menopausal Health Resources
- Clinician Arm (No Intervention): Clinicians were consented in order to have their clinic visits audio recorded. No outcomes data were collected from clinician participants.

INTERVENTIONS:
Behavioral: Starting the Conversation Video — The Starting the Conversation program is designed to increase self-efficacy and outcome expectancies for communicating with providers about sexual health and related issues, reduce barriers to communication, and provide basic training in skills for communicating with providers about these topics, including prioritizing concerns, tips for effective communication, communication practice, and self-feedback.
  Arms: Resources + Video
Behavioral: Sexual and Menopausal Health Resources — Patients will receive a resource list that includes both web-based resources on menopausal and sexual health and center-specific resources, such as contact information for a menopausal & sexual health clinic.
  Arms: Resources + Video; Resources Only

SUMMARY:
The goal of this study is to evaluate an educational video intervention (called Starting the Conversation) aimed to enhance breast cancer patients' beliefs about and communication with respect to sexual concerns. In the current study, 128 breast cancer outpatients will be randomized to either participate in the video intervention and to receive a resource guide addressing sexual and menopausal health or to receive the resource guide alone. Patients will be asked to participate in the video and/or read through the resource guide prior to their clinic visit with their breast cancer provider. The investigators will examine effects of the interventions on patients' beliefs about communication about sexual health and on patients' communication about sexual health during clinic visits with their providers. Secondarily, the investigators will examine effects of the interventions on sexual outcomes and other health outcomes, including psychological well-being and health-related QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving any treatment for breast cancer or have completed acute treatment for breast cancer < 10 years ago
2. Attending clinic visits in the course of follow-up care (i.e., not an initial consult visit)
3. Willing to have clinic visit audio recorded

Exclusion Criteria:

1. Unable to speak English
2. Eastern Cooperative Oncology Group (ECOG) Performance score > 2 OR too ill to participate as judged by physician, self-report, or observation of the research team member
3. Overt cognitive dysfunction or psychiatric disturbance or severe mental illness (e.g., dementia, suicidal behavior, or psychosis), as observed or judged by the researcher or referring source.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-05-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants complete consent and baseline survey before being assigned to a study group.
Groups:
- Clinician Arm: Clinicians were consented in order to have their clinic visits audio recorded. Outcomes data were not collected from clinician participants.
Period: Overall Study
Arm/Group | Resources Only | Resources + Video | Clinician Arm
Started | 71 | 73 | 9
Completed | 69 | 71 | 9
Not Completed | 2 | 2 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinician Arm: Clinicians were consented in order to have their clinic visits audio recorded. Outcomes data was not collected from clinician participants.
- Total: Total of all reporting groups
Arm/Group | Resources Only | Resources + Video | Clinician Arm | Total
Number analyzed (Participants) | 71 | 73 | 9 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  years
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 56.1 (10.9) | 55.8 (11.2) |  | 56.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Female | 71 | 73 |  | 144
    Male | 0 | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Hispanic or Latino | 3 | 3 |  | 6
    Not Hispanic or Latino | 68 | 70 |  | 138
    Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    American Indian or Alaska Native | 0 | 0 |  | 0
    Asian | 0 | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Black or African American | 13 | 26 |  | 39
    White | 53 | 43 |  | 96
    More than one race | 3 | 1 |  | 4
    Unknown or Not Reported | 2 | 3 |  | 5
Months Since Breast Cancer Diagnosis [Mean (Standard Deviation); unit: months] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  months
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 56.6 (64.4) | 43.8 (42.6) |  | 50.12 (54.64)
Relationship Status [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    In a romantic relationship | 46 | 51 |  | 97
    Not in a romantic relationship | 25 | 22 |  | 47
Education Level [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Some high school | 2 | 2 |  | 4
    High school or GED | 12 | 12 |  | 24
    Some college | 17 | 22 |  | 39
    Completed college/graduate school | 40 | 37 |  | 77
Employment Status [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Full or part time | 39 | 40 |  | 79
    Retired | 18 | 15 |  | 33
    Unemployed/disability/other | 14 | 18 |  | 32
Sexual Orientation [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Heterosexual/straight | 70 | 70 |  | 140
    Homosexual/lesbian | 1 | 2 |  | 3
    Bisexual | 0 | 1 |  | 1
Menopausal Status [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Pre-menopausal/peri-menopausal | 18 | 20 |  | 38
    Post-menopausal | 53 | 53 |  | 106
Breast Cancer Stage [Count of Participants; unit: Participants] — Breast cancer stage was assigned by their oncologist using AJCC 7th and 8th edition staging criteria, with stage I having the best prognosis and stage IV having the worst prognosis. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Stage I | 35 | 31 |  | 66
    Stage II | 18 | 23 |  | 41
    Stage III | 8 | 8 |  | 16
    Stage IV | 10 | 11 |  | 21
Surgery Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Breast conserving (lumpectomy) | 43 | 40 |  | 83
    Mastectomy with reconstruction | 23 | 23 |  | 46
    Mastectomy without reconstruction | 2 | 7 |  | 9
    No surgery | 3 | 3 |  | 6
Chemotherapy Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Received chemotherapy | 44 | 51 |  | 95
    No chemotherapy | 27 | 22 |  | 49
Endocrine Therapy Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Received endocrine therapy | 57 | 50 |  | 107
    No endocrine therapy | 14 | 23 |  | 37
Ovarian Suppression Therapy Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Ovarian suppression therapy received | 4 | 4 |  | 8
    No ovarian suppression therapy | 67 | 69 |  | 136
Radiation Therapy Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Radiation received | 48 | 44 |  | 92
    No radiation | 23 | 29 |  | 52
Immunotherapy Received [Count of Participants; unit: Participants] — Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Immunotherapy received | 26 | 22 |  | 48
    No immunotherapy | 45 | 51 |  | 96
Self-Efficacy for Communicating About Sexual Health Issues [Mean (Standard Deviation); unit: score on a scale] — Two items assessed patients' self-efficacy (confidence) for communicating with their breast cancer clinician about sexual health concerns in terms of either talking (item 1) or asking (item 2) about sexual health. Response options used an 11-point scale (0=not at all confident/not at all to 10=extremely confident/very much). Mean scores across the two items were used, ranging from 0-10. Higher scores indicate higher self-efficacy. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 7.7 (2.4) | 7.4 (2.6) |  | 7.5 (2.5)
Outcome Expectancies for Communicating About Sexual Health Issues [Mean (Standard Deviation); unit: score on a scale] — Five items assessed the belief that discussing sexual health with her breast cancer clinician would lead to positive outcomes (e.g., "find a solution to a problem"). Response options used an 11-point scale (0=not at all to 10=very much). Mean scores across the five items were used, ranging from 0-10. Higher scores indicate higher expectancies for positive outcomes. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 7.6 (2.4) | 7.4 (2.6) |  | 7.5 (2.4)
Sexual Function [Mean (Standard Deviation); unit: t-score] — Sexual function was assessed using the Lubrication, Vaginal Discomfort, Satisfaction, and Interest domain scores from the PROMIS SexFS Brief Profile Version 2.0. Higher scores for all domains except Vaginal Discomfort signify better function. Scores are converted to a T-score metric where a score of 50 equates to the mean of the U.S. population of sexually active adults (SD=10). Population: The sexual interest item was administered to all participants, and the lubrication, vaginal discomfort, and satisfaction items were only administered to participants who reported being sexually active. Baseline/outcomes data was not analyzed from clinician participants (N=9)
  t-score
    Vaginal lubrication: number analyzed (Participants) | 35 | 41 | 0 | 76
    Vaginal lubrication | 42.8 (10.1) | 41.6 (8.1) |  | 42.2 (9.0)
    Vaginal discomfort: number analyzed (Participants) | 35 | 41 | 0 | 76
    Vaginal discomfort | 56.1 (10.7) | 58.0 (11.1) |  | 57.2 (10.9)
    Sexual satisfaction: number analyzed (Participants) | 35 | 41 | 0 | 76
    Sexual satisfaction | 46.3 (8.1) | 46.0 (9.1) |  | 46.2 (8.6)
    Sexual interest: number analyzed (Participants) | 71 | 73 | 0 | 144
    Sexual interest | 35.6 (9.9) | 36.6 (11.9) |  | 36.1 (11.0)
General Self-Efficacy for Communication With Provider [Mean (Standard Deviation); unit: score on a scale] — Patients' self-efficacy for communicating with provider generally, as measured through the Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5). The PEPPI-5 is a five-item scale that measures patient confidence in communicating with providers. Response options are on a scale from 1 (Not at All Confident) to 5 (Very Confident) and are summed for a total self-efficacy score (Range: 5-25). Higher scores indicate higher self-efficacy. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 21.6 (3.4) | 21.1 (3.4) |  | 21.3 (3.4)
Barriers to Communicating About Sexual Health [Mean (Standard Deviation); unit: score on a scale] — Patient barriers to communication about sexual health, as measured through a 13-item scale. Scale items cover potential reasons a patient might not want to discuss sexual health concerns with her provider (e.g., "I might become embarrassed"). Items are scored on a 1-5 scale where 1=Strongly Disagree and 5=Strongly Disagree and are summed for a total Barrier score (Range: 13-65). Higher scores indicate more perceived barriers to communication. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 29.6 (8.9) | 30.5 (9.9) |  | 30.1 (9.4)
Patient Anxiety [Mean (Standard Deviation); unit: score on a scale] — Patients self-reported anxiety, as measured through anxiety subscale of the Hospital Anxiety & Depression Scale (HADS). The anxiety subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of anxiety. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 7.3 (4.2) | 7.5 (4.6) |  | 7.4 (4.4)
Patient Depression [Mean (Standard Deviation); unit: score on a scale] — Patients self-reported depression, as measured through depression subscale of the Hospital Anxiety & Depression Scale (HADS). The depression subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of depression. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 4.4 (3.4) | 5.3 (4.0) |  | 4.9 (3.7)
Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Quality of life, as measured through the Abbreviated Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) total score. The FACT-B contains 23 items about physical, functional, and emotional well-being in the context of breast cancer. Scale items are scored from 0 to 4. Summed scores run from 0 to 92, with higher scores indicating higher quality of life. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  score on a scale
    number analyzed (Participants) | 71 | 73 | 0 | 144
    (all) | 61.9 (14.3) | 60.8 (16.7) |  | 61.3 (15.5)
Sexual Activity [Count of Participants; unit: Participants] — Sexual activity was measured by a single item asking (yes/no) whether the participant had any kind of sexual activity in the past 30 days. Population: Baseline/outcomes data was not analyzed from clinician participants (N=9)
  Participants
    number analyzed (Participants) | 71 | 73 | 0 | 144
    Sexually active | 35 | 41 |  | 76
    Not sexually active | 35 | 32 |  | 67
    Refused to answer | 1 | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Self-Efficacy for Communicating About Sexual Health Issues
Description: Two items assessed patients' self-efficacy (confidence) for communicating with their breast cancer clinician about sexual health concerns in terms of either talking (item 1) or asking (item 2) about sexual health. Response options used an 11-point scale (0=not at all confident/not at all to 10=extremely confident/very much). Mean scores across the two items were used, ranging from 0-10. Higher scores indicate higher self-efficacy.
Time Frame: 2 weeks
Population: All participants in the Resources Only arm and 71/73 participants in the Resources + Video arm completed this measure at 2 weeks. Two participants in the Resources + Video arm withdrew from the study before the 2-week assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 8.5 (1.8) | 8.8 (2.1)

2. Primary Outcome: Self-Reported Self-Efficacy for Communicating About Sexual Health Issues
Description: as for outcome 1
Time Frame: 2 months
Population: 69/71 participants in the Resources Only arm and 71/73 participants in the Resources + Video arm completed this measure at 2 months. Two participants in the Resources + Video arm withdrew from the study before the 2-week assessment, and two participants in the Resources Only arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 7.8 (2.0) | 8.2 (2.2)

3. Primary Outcome: Self-Reported Outcome Expectancies for Sexual Health Communication
Description: Five items assessed the belief that discussing sexual health with her breast cancer clinician would lead to positive outcomes (e.g., "find a solution to a problem"). Response options used an 11-point scale (0=not at all to 10=very much). Mean scores across the five items were used, ranging from 0-10. Higher scores indicate higher expectancies for positive outcomes.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 8.2 (2.2) | 8.4 (2.0)

4. Primary Outcome: Self-Reported Outcome Expectancies for Sexual Health Communication
Description: as for outcome 3
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 7.8 (2.1) | 7.8 (2.2)

5. Primary Outcome: Number of Patients Who Asked at Least One Question About Sexual Health at Their Clinic Visit
Description: As coded from clinic visit audio, the number of patients who ask at least one question about sexual health.
Time Frame: 2 weeks
Population: 64/71 participants in the Resources Only arm and 63/73 participants in the Resources + Video arm had their clinic encounters audio recorded and coded. Common reasons why encounters were not recorded include scheduling issues (patient canceled/rescheduled her appointment or attended at a time when recorders were not available) and patient being seen by a non-participating provider (i.e., a provider that did not agree to have their visits audio recorded).
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 64 | 63
Participants | 12 | 25

6. Primary Outcome: Number of Patients Who Initiate Conversation About Sexual Health in Their Clinic Visit
Description: As coded from clinic visit audio, the number of patients who raise the topic of sexual health during their encounter (out of encounters where a sexual health discussion occurred).
Time Frame: 2 weeks
Population: Encounters where the provider raised the topic of sexual health were excluded from this analysis, as it is not known whether the patient would have raised the topic had the provider not raised it first.
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 47 | 39
Participants | 14 | 20

7. Secondary Outcome: Recruitment Rates (Feasibility)
Description: Recruitment rates, as measured by percentage of patients enrolled (i.e., baselined) out of eligible patients approached for the study.
Time Frame: baseline
Population: 177 eligible candidates were approached for participation in the intervention trial.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Recruitment rates are calculated for all potential study candidates.
Arm/Group | All Participants
Number analyzed (Participants) | 177
Participants | 144

8. Secondary Outcome: Retention Rates (Feasibility)
Description: Retention rates, as measured by percentage of patients who remain on study for 2-week follow-up assessment.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 73
Participants | 71 | 71

9. Secondary Outcome: Retention Rates (Feasibility)
Description: Retention rates, as measured by percentage of patients who remain on study for 2-month follow-up assessment.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 73
Participants | 69 | 71

10. Secondary Outcome: Intervention Acceptability
Description: Acceptability of intervention, as measured through the item "Overall, how satisfied were you with this program?". Responses options include Very Satisfied, Satisfied, Dissatisfied, and Very Dissatisfied. Responses of "satisfied" or "very satisfied" indicate acceptability. Number of patients reporting acceptability and number of patients not reporting acceptability are presented.
Time Frame: 2 weeks
Population: Participants who did not complete the intervention (i.e., reported not watching the vide) and did not complete the 2-week survey were not administered this item. 64/73 participants both completed the intervention and the 2-week follow-up survey.
Measure: Count of Participants; unit: Participants
Groups:
- Resources + Video Group Only: Patients will receive a list of web resources on sexual and menopausal health in breast cancer. In addition to the resources, patients will be asked to view an online video called "Starting the Conversation" and to complete an accompanying workbook. Patients in this arm will be asked to review the resource list, watch the Starting the Conversation video, and complete the workbook before their next clinic visit.
  Starting the Conversation Video: The Starting the Conversation program is designed to increase self-efficacy and outcome expectancies for communicating with providers about sexual health and related issues, reduce barriers to communication, and provide basic training in skills for communicating with providers about these topics, including prioritizing concerns, tips for effective communication, communication practice, and self-feedback.
  Sexual and Menopausal Health Resources: Patients will receive a resource list that includes both web-based resources on menopausal and sexual health and center-specific resources, such as contact information for a menopausal & sexual health clinic.
Arm/Group | Resources + Video Group Only
Number analyzed (Participants) | 64
Participants
  Satisfied/Very Satisfied | 64
  Dissatisfied/Very Dissatisfied | 0

11. Secondary Outcome: Sexual Activity
Description: Sexual activity was measured by a single item asking (yes/no) whether the participant had any kind of sexual activity in the past 30 days.
Time Frame: 2 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
Participants
  Sexually active | 32 | 50
  Not sexually active | 37 | 21

12. Secondary Outcome: Sexual Function
Description: Sexual function was assessed using the Lubrication, Vaginal Discomfort, Satisfaction, and Interest domain scores from the Patient-Reported Outcomes Measurement Information System Sexual Function and Satisfaction scale (PROMIS SexFS) Brief Profile Version 2.0. Scores are converted to a T-score metric where a score of 50 equates to the mean of the U.S. population of sexually active adults (SD=10). Higher scores for all domains except Vaginal Discomfort signify better function.
Time Frame: 2 months
Population: 69/71 Resources Only and 71/73 Resources + Video participants completed the 2-month follow-up. Only participants who reported being sexually active in the past month were given the items regarding vaginal lubrication, vaginal discomfort, and sexual satisfaction (32/69 Resources Only patients and 50/71 Resources + Video patients). All participants were given the item on sexual interest.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
t-score
  Vaginal lubrication: number analyzed (Participants) | 32 | 50
  Vaginal lubrication | 42.2 (8.5) | 41.6 (9.7)
  Vaginal discomfort: number analyzed (Participants) | 32 | 50
  Vaginal discomfort | 55.8 (11.8) | 58.4 (11.1)
  Sexual satisfaction: number analyzed (Participants) | 32 | 50
  Sexual satisfaction | 44.7 (7.3) | 46.3 (8.5)
  Sexual interest | 35.7 (9.7) | 37.8 (11.2)

13. Secondary Outcome: General Self-Efficacy for Communication With Provider
Description: Patients' self-efficacy for communicating with provider generally, as measured through the Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5). The PEPPI-5 is a five-item scale that measures patient confidence in communicating with providers. Response options are on a scale from 1 (Not at All Confident) to 5 (Very Confident) and are summed for a total self-efficacy score (Range: 5-25). Higher scores indicate higher self-efficacy.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 21.6 (3.5) | 22.2 (3.0)

14. Secondary Outcome: Barriers to Communicating About Sexual Health
Description: Patient barriers to communication about sexual health, as measured through a 13-item scale. Scale items cover potential reasons a patient might not want to discuss sexual health concerns with her provider (e.g., "I might become embarrassed"). Items are scored on a 1-5 scale where 1=Strongly Disagree and 5=Strongly Disagree. A total barrier score will be taken from this scale (Range: 13-65). Higher scores indicate more perceived barriers to communication.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 29.0 (9.0) | 27.8 (9.9)

15. Secondary Outcome: Self-Reported Anxiety
Description: Patients self-reported anxiety, as measured through anxiety subscale of the Hospital Anxiety & Depression Scale (HADS). The anxiety subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 7.3 (4.2) | 6.6 (4.9)

16. Secondary Outcome: Self-Reported Depression
Description: Patients self-reported depression, as measured through depression subscale of the Hospital Anxiety & Depression Scale (HADS). The depression subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of depression.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 4.4 (3.5) | 4.6 (3.7)

17. Secondary Outcome: Self-Reported Quality of Life
Description: Quality of life, as measured through the Abbreviated Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) total score. The FACT-B contains 23 items about physical, functional, and emotional well-being in the context of breast cancer. Scale items are scored from 0 to 4. Summed scores run from 0 to 92, with higher scores indicating higher quality of life.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 62.6 (13.9) | 61.8 (18.2)

18. Secondary Outcome: Self-Reported Self-Efficacy for Communicating About About Treatment Side Effects
Description: Patients' self-reported self-efficacy for communication about treatment side effects with their breast cancer provider. The items about treatment side effects consist of 2 items within a larger 6-item scale which ask the patient how confident she is in talking to her provider about treatment side effects and asking her provider about treatment side effects. Response options range from 0 (not at all confident) to 10 (extremely confident). Mean scores will be reported.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 9.3 (1.5) | 9.5 (1.3)

19. Secondary Outcome: Self-Reported Self-Efficacy for Communicating About About Treatment Side Effects
Description: as for outcome 18
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 9.1 (1.3) | 9.3 (1.2)

20. Secondary Outcome: Self-Reported Self-Efficacy for Communicating About About Menopausal Health
Description: Patients' self-reported self-efficacy for communication about menopausal health with their breast cancer provider. The items about menopausal health consist of 2 items within a larger 6-item scale which ask the patient how confident she is in talking to her provider about menopausal health and asking her provider about menopausal health. Response options range from 0 (not at all confident) to 10 (extremely confident). Mean scores will be reported.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 9.1 (1.6) | 9.4 (1.5)

21. Secondary Outcome: Self-Reported Self-Efficacy for Communicating About About Menopausal Health
Description: as for outcome 20
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 9.0 (1.4) | 9.3 (1.2)

22. Secondary Outcome: Self-Reported Outcome Expectancies for Communication About Treatment Side Effects
Description: Five items assessed the belief that discussing treatment side effects with her breast cancer clinician would lead to positive outcomes (e.g., "find a solution to a problem"). Response options used an 11-point scale (0=not at all to 10=very much). Mean scores across the five items were used, ranging from 0-10. Higher scores indicate higher expectancies for positive outcomes.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 8.9 (1.4) | 9.2 (1.2)

23. Secondary Outcome: Self-Reported Outcome Expectancies for Communication About Treatment Side Effects
Description: as for outcome 22
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 8.6 (1.5) | 8.8 (1.4)

24. Secondary Outcome: Self-Reported Outcome Expectancies for Communication About Menopausal Health
Description: Five items assessed the belief that discussing menopausal health with her breast cancer clinician would lead to positive outcomes (e.g., "find a solution to a problem"). Response options used an 11-point scale (0=not at all to 10=very much). Mean scores across the five items were used, ranging from 0-10. Higher scores indicate higher expectancies for positive outcomes.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 71 | 71
score on a scale | 8.6 (1.7) | 8.7 (2.0)

25. Secondary Outcome: Self-Reported Outcome Expectancies for Communication About Menopausal Health
Description: as for outcome 24
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Only | Resources + Video
Number analyzed (Participants) | 69 | 71
score on a scale | 8.3 (1.8) | 8.7 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 2 months.
Description: An adverse event is defined as a distress reaction during any study event, including survey completion and intervention participation.
Groups:
- Clinician Arm: Clinicians were consented in order to have their clinic visits audio recorded.
Arm/Group | Resources Only | Resources + Video | Clinician Arm
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73 | 0/9
Other Adverse Events (participants affected / at risk) | 0/71 | 0/73 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03624972/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03624972/ICF_003.pdf